CLINICAL TRIAL: NCT04986735
Title: Evaluation of Safety and Efficacy of Empagliflozin for Neutropenia and Neutrophil Dysfunction in Children With Glycogen Storage Disease Type 1b (GSD1b)
Brief Title: Prospective Cohort Study of Children With GSD1b Receiving Empagliflozin
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hong Kong Children's Hospital (Other)
Responsible Party: Principal Investigator, Kwok Mei-kwun, Associate Consultant, Hong Kong Children's Hospital
Other Study IDs: KWOK-HKCH-GSD1-EMPA
Record Dates: First submitted 2021-07-27; First posted 2021-08-03 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Glycogen Storage Disease Type IB
MeSH Terms: conditions — Glycogen Storage Disease IB | interventions — empagliflozin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Empagliflozin — All subjects will have a baseline assessment and be prospectively followed up for 52 weeks to examine their outcome after receiving empagliflozin for neutropenia and neutrophil dysfunction.
  Other Names: Jardiance

SUMMARY:
This is a prospective cohort study of children with GSD1b to evaluate their outcome after using empagliflozin for neutrophil defects.

DETAILED DESCRIPTION:
Glycogen Storage Disease Type 1b (GSD1b) is an ultra-rare inborn error of carbohydrate metabolism, characterized by low neutrophil count, neutrophil dysfunction, and the associated recurrent infections and inflammatory bowel conditions.

The current standard treatment with granulocyte colony-stimulating factor (GCSF) only increases neutrophil count but does not improve neutrophil function. It achieves only partial clinical response. Fever, recurrent infections, and gastrointestinal upset remain significant problems. Long-term regular GCSF injection is needed to sustain the clinical effect, but is also associated with development of serious complications including massive spleen enlargement, acute myeloid leukemia and myelodysplastic syndrome.

Accumulation of a toxic metabolite called 1,5-anhydroglucitol-6-phosphate (1,5AG6P) is recently discovered as the cause of neutrophil problems in GSD1b. Empagliflozin, a sodium-glucose co-transporter 2 (SGLT2) inhibitor widely used as anti-diabetic drug, is known to promote excretion of 1,5-anhydroglucitol (1,5AG) in kidney. Since 1,5AG is the precursor of 1,5AG6P, empagliflozin also reduces the accumulation of 1,5AG6P. This is confirmed by animal studies that empagliflozin is shown to improve neutrophil count and function in GSD1b mouse model. Similar benefits are also recently reported in human cases (3 adults and 2 children with GSD1b), that GCSF dose could be significantly reduced or even stopped.

This is a prospective cohort study of children with GSD1b to examine their outcome after receiving empagliflozin treatment. The objective is to evaluate the short to medium term safety and efficacy of empagliflozin. The ultimate goal is to assess if SGLT2 inhibitor could be an effective alternative of GCSF with less side effects and risks, and to improve the clinical outcomes and quality of life for patients and families with GSD1b.

ELIGIBILITY:
Inclusion Criteria:

- Subject (aged 6 months to 18 years) is enzymatically/genetically confirmed to have GSD 1b and has been on regular GCSF treatment for >= 1 month

Exclusion Criteria:

* Subject fails to provide relevant background medical information, or comply with all requirements of the clinical trial, or sign the informed consent
* Subject has any co-morbidity or condition that could increase the risk of empagliflozin treatment (e.g. renal failure with eGFR <30 mL/min/1.73m2 or requiring dialysis, diabetes requiring insulin &/or oral hypoglycemic agents, dyslipidemia requiring pharmacological intervention)
* Subject is pregnant, or a sexually active female who does not consent to use effective contraception during the study
* History of liver transplantation is NOT an exclusion criterium

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: GSD 1b patients (aged 6 months to 18 years) with diagnosis confirmed by enzymatic and/or genetic analysis, and has been on regular GCSF treatment for >= 1 month
Sampling Method: Probability Sample
Enrollment: 11 (Estimated)
Dates: Start 2021-08-08 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of empagliflozin - usage of granulocyte colony stimulating factor (GCSF) | from the start to the 52nd week of empagliflozin treatment
  Dosage and frequency of administration of GCSF

SECONDARY OUTCOMES:
Efficacy of empagliflozin - neutrophil number and function | from the start to the 52nd week of empagliflozin treatment
  Average neutrophil count and neutrophil oxidative burst
Efficacy of empagliflozin - bowel manifestations | from the start to the 52nd week of empagliflozin treatment
  Severity of bowel inflammation, diarrhea, and aphthous ulcers
Efficacy of empagliflozin - frequency of infections | from the start to the 52nd week of empagliflozin treatment
  Number of infections requiring hospitalization and antibiotics/surgical intervention
Efficacy of empagliflozin - biochemical improvement | from the start to the 52nd week of empagliflozin treatment
  Blood 1,5-anhydroglucitol level and urine glucose excretion
General metabolic control - GSD1b metabolic & imaging profile, concomitant interventions | from the start to the 52nd week of empagliflozin treatment
  Metabolic profile and concomitant interventions that reflects metabolic control of GSD1b
General well being - Quality of life | from the start to the 52nd week of empagliflozin treatment
  Pediatric Quality of Life Inventory™ (PedsQL™) - English or Cantonese/Chinese versions
Safety of empagliflozin - presence or absence of hypoglycemia | from the start to the 52nd week of empagliflozin treatment
  Frequency of symptomatic or severe hypoglycemia, average glucose levels
Safety of empagliflozin - prescence of absence of empagliflozin-related side effects | from the start to the 52nd week of empagliflozin treatment
  number of empagliflozin-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Mei Kwun Kwok, Principal Investigator — Hong Kong Children's Hospital
Locations (1):
- Hong Kong Children's Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No